CLINICAL TRIAL: NCT01769365
Title: Comparison of 7-day Triple, 10-day Sequential, and 7-day Concomitant Therapies for Helicobacter Pylori Infection in Taiwan
Brief Title: Concomitant, Sequential, and Standard Triple Therapy for H. Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Chief of Division of Gastroenterology; Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS99-CT7-10
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2015-10-06 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2015-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori infection
MeSH Terms: interventions — Pantoprazole; Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 7-day quadruple therapy (Experimental): 1. pantoprazole 40 mg twice daily for 7 days,
  2. clarithromycin 500 mg twice daily for 7 days,
  3. amoxicillin 1 g twice daily for 7 days,
  4. metronidazole 500 mg twice daily for 7 days
  Interventions: Drug: 7-day quadruple therapy
- 10-day sequential therapy (Experimental): 1. pantoprazole 40 mg twice daily for 5 days and amoxicillin 1 g twice daily for 5 days, followed by
  2. pantoprazole 40 mg twice daily for 5 days, clarithromycin 500 mg twice daily for 5 days, metronidazole 500 mg twice daily for 5 days.
  Interventions: Drug: 10-day sequential therapy
- 7-day standard triple therapy (Active Comparator): 1. pantoprazole 40 mg twice daily for 7 days,
  2. clarithromycin 500 mg twice daily for 7 days,
  3. amoxicillin 1 g twice daily for 7 days.
  Interventions: Drug: 7-day standard triple therapy

INTERVENTIONS:
Drug: 7-day quadruple therapy — pantoprazole 40 mg twice daily, clarithromycin 500 mg twice daily, amoxicillin 1 g twice daily and metronidazole 500 mg twice daily for 7 days
  Other Names: Pantoprazole, amoxicillin, clarithromycin, metronidazole
  Arms: 7-day quadruple therapy
Drug: 10-day sequential therapy — pantoprazole 40 mg twice daily and amoxicillin 1 g twice daily for 5 days, followed by pantoprazole 40 mg twice daily, clarithromycin 500 mg twice daily and metronidazole 500 mg twice daily for a further 5 days
  Other Names: sequential group
  Arms: 10-day sequential therapy
Drug: 7-day standard triple therapy — pantoprazole 40 mg twice daily, clarithromycin 500 mg twice daily, and amoxicillin 1 g twice daily for 7 days
  Other Names: pantoprazole, clarithromycin, amoxicillin
  Arms: 7-day standard triple therapy

SUMMARY:
To simultaneously compare the efficacies of 7-day triple, 10-day sequential and 7-day quadruple therapies for H. pylori infection in Taiwan. Consecutive H. pylori-infected patients were randomly assigned to a 7-day standard triple therapy (pantoprazole, clarithromycin, and amoxicillin for 7 days), a 10-day sequential therapy (pantoprazole and amoxicillin for 5 days, followed by pantoprazole, clarithromycin and metronidazole for a further 5 days) or a 7-day quadruple therapy (pantoprazole, clarithromycin, amoxicillin and metronidazole for 7 days). The end point is to evaluate the effectiveness of Helicobacter pylori eradication rates between three groups.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of three H. pylori eradication regimens: 7-day standard triple therapy (pantoprazole, clarithromycin, and amoxicillin for 7 days), 10-day sequential therapy (pantoprazole and amoxicillin for 5 days, followed by pantoprazole, clarithromycin and metronidazole for a further 5 days) and 7-day quadruple therapy (pantoprazole, clarithromycin, amoxicillin and metronidazole for 7 days) in Taiwan.

A total of 306 subjects are enrolled into this study.

H. pylori-infected patients are randomized to a 7-day standard triple therapy, a 10-day sequential therapy, or a 7-day quadruple therapy. Eradication efficacy is assessed by a follow-up endoscopy with rapid urease test and histological examination eight weeks after the H. pylori therapy. The eradication rates of three groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive H. pylori-infected outpatients, at least 20 years of age, with endoscopically proven peptic ulcer diseases or gastritis

Exclusion Criteria:

* previous H. pylori-eradication therapy
* ingestion of antibiotics, bismuth, or proton pump inhibitors within the prior 4 weeks
* patients with allergic history to the medications used
* patients with previous gastric surgery
* the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia)
* pregnant women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-I Hsu, MD, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Hsu PI, Wu DC, Chen WC, Tseng HH, Yu HC, Wang HM, Kao SS, Lai KH, Chen A, Tsay FW. Randomized controlled trial comparing 7-day triple, 10-day sequential, and 7-day concomitant therapies for Helicobacter pylori infection. Antimicrob Agents Chemother. 2014 Oct;58(10):5936-42. doi: 10.1128/AAC.02922-14. Epub 2014 Jul 28. PMID 25070099

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We surveyed patients who visited the gastroenterological clinic of Kaohsiung Medical University Hospital (KMUH), Kaohsiung Veteran General Hospital (KVGH). A total of 307 H. pylori-infected patients were randomly assigned to triple (n=103 ) or sequential (n = 102) or concomitant (n = 102) therapies.
Period: Overall Study
Arm/Group | 7-day Quadruple Therapy | 10-day Sequential Therapy | 7-day Standard Triple Therapy
Started | 102 | 102 | 103
Completed | 102 | 100 | 101
Not Completed | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 7-day Quadruple Therapy | 10-day Sequential Therapy | 7-day Standard Triple Therapy | Total
Number analyzed (Participants) | 102 | 102 | 103 | 307
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 74 | 68 | 69 | 211
  >=65 years | 28 | 34 | 34 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.85 (12.31) | 54.96 (12.00) | 56.08 (14.00) | 54.88 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 50 | 41 | 132
  Male | 61 | 52 | 62 | 175
Region of Enrollment [Number; unit: participants]
  Taiwan | 102 | 102 | 103 | 307

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Eradication of Helicobacter Pylori
Description: Evaluate eradication outcome by endoscopy urease test and histology or urea breath test
Time Frame: at the 6th week after the end of anti- H. pylori therapy
Measure: Number; unit: participants
Arm/Group | 7-day Quadruple Therapy | 10-day Sequential Therapy | 7-day Standard Triple Therapy
Number analyzed (Participants) | 102 | 102 | 103
participants | 102 | 100 | 101

ADVERSE EVENTS:
Arm/Group | 7-day Quadruple Therapy | 10-day Sequential Therapy | 7-day Standard Triple Therapy
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/102 | 0/103
Other Adverse Events (participants affected / at risk) | 14/102 | 9/102 | 9/103
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7-day Quadruple Therapy (N=102) | 10-day Sequential Therapy (N=102) | 7-day Standard Triple Therapy (N=103)
Nausea (Gastrointestinal disorders) | 7 (7) | 5 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 7 (7) | 4 (4) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
The trial was performed in a single country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes